CLINICAL TRIAL: NCT03666338
Title: Influence of the Initial Level of Consciousness on Early, Goal-directed Mobilization
Acronym: SOMS-GCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Massachusetts General Hospital (Other); Università degli Studi di Brescia (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Stefan Schaller, Specialist Intensive Care, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOMS-GCS
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Critical Care; Rehabilitation
Keywords: early mobilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early, goal-directed mobilization (Active Comparator): Early goal-directed mobilization with (1) SOMS algorithm and (2) facilitator
  Interventions: Other: Early, goal-directed mobilization
- Standard of Care (No Intervention): Standard of Care regarding mobilization

INTERVENTIONS:
Other: Early, goal-directed mobilization — Early, goal directed mobilization using (1) the SOMS algorithm and (2) facilitator
  Arms: Early, goal-directed mobilization

SUMMARY:
Analysis of the randomized controlled SOMS trial of early, goal-directed mobilization to investigate if the treatment effect is consistent and independent of the initial conscious state without evidence of moderation or modification.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* mechanically ventilated for less than 48 h and expected to require mechanical ventilation for at least another 24 h at the time of screening
* functionally independent at baseline with a Barthel Index Score of at least 70 at 2 weeks before admission to the ICU based on patient or proxy completion of the measure

Exclusion Criteria:

* admitted to hospital for more than 5 days before screening
* a motor component of Glasgow Coma Scale (GCS) lower than 5
* irreversible disorder with a 6-month mortality of greater than 50%,
* raised intracranial pressure
* cardiopulmonary arrest
* unstable fractures contributing to probable immobility
* inclusion in another trial at the same time
* acute myocardial infarction
* do not have lower part of their legs
* have a rapidly developing neuromuscluar disease
* pregnant
* ruptured or leaking aortic aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2015-11-04 (Actual); Study Completion 2016-02-04 (Actual)

PRIMARY OUTCOMES:
Functional independence at hospital discharge | At the day of hospital discharge, on average up to 1 month
  minimal modified functional independence measure score of 8 (Scale ranging from 0-8 with the subdomain locomotion and transfer 0-4 each)

SECONDARY OUTCOMES:
average achieved mobility level during the ICU stay | from ICU admission to ICU discharge, on average up to 2 weeks
  mean achieved SOMS level
Functional status at hospital discharge | At the day of hospital discharge, on average up to 1 month
  minimal modified functional independence measure score (range 0-8) of the subdomains transfer and locomotion with 0-4 each
Start to mobilization (SOMS > 0) | Days from ICU admission till first mobilization, approximately up to 5 days
  Start to mobilization in days (Surgical Optimal Mobilization Scale > 0, ranging from 0 = no mobilization to 4 ambulation)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
On reasonable request from researchers after an agreement has been found.

REFERENCES:
- [Background] Schaller SJ, Anstey M, Blobner M, Edrich T, Grabitz SD, Gradwohl-Matis I, Heim M, Houle T, Kurth T, Latronico N, Lee J, Meyer MJ, Peponis T, Talmor D, Velmahos GC, Waak K, Walz JM, Zafonte R, Eikermann M; International Early SOMS-guided Mobilization Research Initiative. Early, goal-directed mobilisation in the surgical intensive care unit: a randomised controlled trial. Lancet. 2016 Oct 1;388(10052):1377-1388. doi: 10.1016/S0140-6736(16)31637-3. PMID 27707496